CLINICAL TRIAL: NCT01321710
Title: Sleep Disruption in New Parents: An Intervention Trial
Brief Title: Sleep Disruption in New Mothers: An Intervention Trial
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOMS Sleep; 2R01NR005345 (NIH)
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-01

CONDITIONS: Pregnancy; Postpartum Period; Sleep Disturbance
Keywords: sleep hygiene; actigraphy; maternal; infant; postpartum period; immunization; acetaminophen
MeSH Terms: conditions — Parasomnias; Sleep Hygiene | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dietary information & standard care (Active Comparator): Mothers in this arm receive dietary information aimed at reducing postpartum sleep disturbance.
  Infants in this arm receive no intervention beyond standard immunization care.
  Interventions: Behavioral: Dietary information
- Sleep hygiene & standard care (Experimental): Mothers in this arm receive a sleep hygiene intervention aimed at improving their postpartum sleep.
  Infants in this arm receive standard immunization care.
  Interventions: Behavioral: Sleep hygiene
- Sleep hygiene & acetaminophen (Experimental): Mothers in this arm receive a sleep hygiene intervention aimed at improving postpartum sleep.
  Infants in this arm receive an acetaminophen intervention (12.5mg per kg infant weight, 1 dose 30 minutes prior to immunization and q4-6h thereafter, for a total of 5 doses) to minimize sleep disturbance following immunization.
  Interventions: Behavioral: Sleep hygiene; Drug: Acetaminophen

INTERVENTIONS:
Behavioral: Sleep hygiene — This intervention consists of behavioral strategies for minimizing maternal arousal and sleep disturbance as a result of night-time infant care. Key components include: infant proximity, low lighting, and noise attenuation.
  It is administered to women during their last month of pregnancy.
  Arms: Sleep hygiene & acetaminophen; Sleep hygiene & standard care
Behavioral: Dietary information — This intervention consists of dietary information aimed at improving postpartum sleep. The recommendations include avoiding alcohol, caffeine, and heavy meals before bed, as well as eating healthy foods.
  Arms: Dietary information & standard care
Drug: Acetaminophen — 51-90mg depending on infant weight (12.5mg per kg infant weight). Administered 30 minutes prior to immunization and q4-6h for a total of 5 doses.
  Arms: Sleep hygiene & acetaminophen

SUMMARY:
The purpose of this study is to test a behavioral intervention to minimize sleep disruption and fatigue in new mothers after the birth of their first infant. This study also tests whether an acetaminophen intervention at the time of an infant's 2-month immunization series improves infant and maternal sleep.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women expecting first singleton birth
* able to speak, read, and write in English
* willing to participate for 3 consecutive days and nights during 36-39 weeks gestation and at 4, 8, and 12 weeks postpartum
* willing to have their infant participate in ankle actigraphy recording of their sleep/wake patterns for 96 hrs at the time of their first immunization

Exclusion Criteria:

* history of affective illness prior to pregnancy
* current use of medications that may alter sleep
* history of a diagnosed sleep disorder such as sleep apnea, nocturnal myoclonus, or narcolepsy
* plan to employ live-in help with child care
* working the night-shift
* multiple pregnancy with twins or more

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A. Lee, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

REFERENCES:
- [Result] Lee KA, Gay CL. Can modifications to the bedroom environment improve the sleep of new parents? Two randomized controlled trials. Res Nurs Health. 2011 Feb;34(1):7-19. doi: 10.1002/nur.20413. Epub 2010 Nov 17. PMID 21243655
- [Result] Goyal D, Gay C, Lee KA. How much does low socioeconomic status increase the risk of prenatal and postpartum depressive symptoms in first-time mothers? Womens Health Issues. 2010 Mar-Apr;20(2):96-104. doi: 10.1016/j.whi.2009.11.003. Epub 2010 Feb 4. PMID 20133153
- [Result] Kennedy HP, Gardiner A, Gay C, Lee KA. Negotiating sleep: a qualitative study of new mothers. J Perinat Neonatal Nurs. 2007 Apr-Jun;21(2):114-22. doi: 10.1097/01.JPN.0000270628.51122.1d. PMID 17505231
- [Derived] Franck L, Gay CL, Lynch M, Lee KA. Infant sleep after immunization: randomized controlled trial of prophylactic acetaminophen. Pediatrics. 2011 Dec;128(6):1100-8. doi: 10.1542/peds.2011-1712. Epub 2011 Nov 28. PMID 22123869

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietary Information & Standard Care: Mothers in this arm receive dietary information aimed at reducing postpartum sleep disturbance.
  Infants in this arm receive standard immunization care.
- Sleep Hygiene & Acetaminophen: Mothers in this arm receive a sleep hygiene intervention aimed at improving postpartum sleep.
  Infants in this arm receive an acetaminophen intervention to minimize sleep disturbance following immunization.
Period: Overall Study
Arm/Group | Dietary Information & Standard Care | Sleep Hygiene & Standard Care | Sleep Hygiene & Acetaminophen
Started | 50 | 58 | 44
Completed | 46 | 53 | 44
Not Completed | 4 | 5 | 0
Not completed — Lost to Follow-up | 4 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietary Information & Standard Care | Sleep Hygiene & Standard Care | Sleep Hygiene & Acetaminophen | Total
Number analyzed (Participants) | 50 | 58 | 44 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 58 | 44 | 152
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.5) | 26.4 (6.4) | 26.5 (7.1) | 26.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 58 | 44 | 152
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 58 | 44 | 152

OUTCOME MEASURES:

1. Primary Outcome: Maternal Sleep Quantity (Objective)
Description: Maternal sleep quantity is defined as total night-time sleep in hours as measured by wrist actigraphy over 3 nights.
Time Frame: 1-month postpartum (approximately)
Population: ITT analysis. Because this was a repeated measures analysis at 1 and 3 months postpartum, subjects missing outcome data at either point were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Dietary Information: Mothers in this group received dietary information for improving sleep.
- Sleep Hygiene: Mothers in this group received sleep hygiene information
Arm/Group | Dietary Information | Sleep Hygiene
Number analyzed (Participants) | 32 | 77
hours | 6.1 (1.4) | 6.6 (1.3)

2. Primary Outcome: Maternal Sleep Quality (Objective)
Description: Maternal sleep quality is defined as sleep efficiency (percent sleep per time in bed averaged across 3 nights) as measured by wrist actigraphy.
Time Frame: 1 month postpartum (approximately)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep per time in bed
Arm/Group | Dietary Information | Sleep Hygiene
Number analyzed (Participants) | 32 | 77
percentage of sleep per time in bed | 68 (11) | 71 (10)

3. Secondary Outcome: Maternal Sleep Disturbance (Subjective)
Description: Maternal sleep disturbance is measured by the total score on the General Sleep Disturbance Scale (GSDS). The GSDS is a self-report questionnaire that measures perceived sleep disturbance in the past week. GSDS scores range from 0 to 147, with higher scores indicating more sleep disturbance.
Time Frame: 1 month postpartum (approximately)
Population: ITT analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dietary Information | Sleep Hygiene
Number analyzed (Participants) | 44 | 92
Scores on a scale | 49.9 (17.9) | 49.4 (14.6)

4. Secondary Outcome: Maternal Well-being
Description: Maternal well-being was measured by the total score on the Center for Epidemiologic Studies - Depression Scale (CES-D). The CES-D measures depressive symptoms in the past week. CES-D scores can range 0 to 60, with higher scores indicating more symptoms of depression.
Time Frame: 1 month postpartum (approximately)
Population: ITT analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dietary Information | Sleep Hygiene
Number analyzed (Participants) | 44 | 91
Scores on a scale | 13.3 (7.7) | 13.0 (7.9)

5. Primary Outcome: Change in Infant Sleep Quantity (Objective)
Description: Change in infant sleep quantity is defined as the difference between the number of hours slept in the 24 hours prior to immunization and the the number of hours slept after immunization (positive numbers indicate more sleep following immunization). Infant sleep was measured by ankle actigraphy.
Time Frame: 24 hours before and 24 hours after immunizations at approximately 2 months of age
Population: ITT analysis. Infants who were not immunized or did not have valid outcome data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Standard Immunization Care: Infants in this group received standard immunization care from their health care provider (may or may not have included prophylactic acetaminophen).
- Prophylactic Acetaminophen: Infants in this group received prophylactic acetaminophen administered prior to immunization and 4 subsequent doses administered in the 24 hours following immunization.
Arm/Group | Standard Immunization Care | Prophylactic Acetaminophen
Number analyzed (Participants) | 21 | 49
minutes | 47.4 (133.3) | 73.1 (151.8)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Dietary Information & Standard Care | Sleep Hygiene & Standard Care | Sleep Hygiene & Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/58 | 0/50
Other Adverse Events (participants affected / at risk) | 0/44 | 0/58 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No